CLINICAL TRIAL: NCT01805596
Title: Effect of Ticagrelor on Endothelial Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ENTC-18129
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease; Endothelial Function
Keywords: coronary artery disease; endothelial function; antiplatelet agent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- clopidogrel-ticagrelor (Experimental): 21 days clopidogrel followed by 21 days ticagrelor
  Interventions: Drug: clopidogrel; Drug: Ticagrelor
- ticagrelor-clopidogrel (Experimental): ticagrelor for 21 days followed by clopidogrel for 21 days
  Interventions: Drug: clopidogrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: clopidogrel
  Other Names: Plavix
Drug: Ticagrelor
  Other Names: Brilinta

SUMMARY:
This study is to assess the function of blood vessels while being treated with different types of blood thinners to determine the effect of these medications on blood vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old
2. At least two cardiovascular risk factors
3. Demonstrated endothelial dysfunction
4. Evidence of coronary artery disease

Exclusion Criteria:

1. Second (II) or third (III) degree heart block without a pacemaker
2. Known active pathological bleeding, history of stroke, or bleeding diathesis
3. Dyspnea classified as NYHA class III-IV
4. Need for oral anticoagulants
5. Clinically significant valvular heart disease
6. Any concurrent life threatening condition with a life expectancy less than 1 year
7. History or evidence of drug or alcohol abuse within the last 12 months
8. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
9. History of hypersensitivity to any of the study drugs or to medications belonging to the same therapeutic class as the study drugs as well as known or suspected contraindications to the study drugs.
10. Latex allergy
11. History of noncompliance to medical regimens or unwillingness to comply with the study protocol
12. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer Positive pregnancy test, breast feeding women or women of child bearing potential not using highly effective methods of contraception.
13. Patients who are also taking strong CYP3A4 inhibitors (e.g., ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir)
14. patients taking antiplatelet medications which cannot be stopped
15. severe liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Endothelial Function after 21 days of antiplatelet medication | 21 days
  The change in endothelial function from baseline will be assessed after 21 days of clopidogrel; the change in endothelial function from baseline will be assessed after 21 days of ticagrelor. This will be measured using RH-PAT units.

SECONDARY OUTCOMES:
Acute change in endothelial function | 2 hours
  Endothelial function assessed 2 hours post ticagrelor

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Alemayehu M, Kim RB, Lavi R, Gong I, D'Alfonso S, Mansell SE, Wall S, Lavi S. Effect of Ticagrelor Versus Clopidogrel on Vascular Reactivity. J Am Coll Cardiol. 2017 May 2;69(17):2246-2248. doi: 10.1016/j.jacc.2017.02.048. No abstract available. PMID 28449783